CLINICAL TRIAL: NCT00407836
Title: Phase II Study of Efficacy, Tolerability and Safety of CD4-Specific T-cell Vaccine in HIV Infection
Brief Title: Efficacy Study of T Cell Vaccination in HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Zvi Bentwich, M.D, Ben Gurion University of the Negev
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sor444006ctil
Record Dates: First submitted 2006-12-03; First posted 2006-12-05 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2006-11

CONDITIONS: HIV Infections
Keywords: HIV; CD4 T cell level; CD4 autoimmunity; Viral load; T cell vaccination; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccination (Experimental): One arm of open label T cell vaccination in which all participants will receive the T cell vaccine
  Interventions: Biological: T cell vaccination

INTERVENTIONS:
Biological: T cell vaccination — Approximately 10-20 million glutaraldehyde fixed CD4 responsive autologous T cells in 1-2 ml, per vaccine injection.
Biological: T cell vaccination — Approximately 10-20 million autologous CD4 reactive T cells per each vaccine injection

SUMMARY:
The hallmark of HIV infection and AIDS is the continuous attrition of CD4 T cells. One of the mechanisms that may account for the CD4 attrition , is autoimmunity against the CD4 T cells, caused by autologous immune cells. Vaccination against autoimmune reactive T cells has been successfully tried in animal models of autoimmune diseases and is now being tried in patients with Multiple Sclerosis. The purpose of the present study is to test this hypothesis in HIV infection. We will vaccinate HIV infected patients in whom specific autoimmune reactivity against CD4 is present , with their own CD4 reactive T cells. Following that, we shall study the patients and find out if the T cell vaccination caused a rise in CD4 T cell levels, and whether it influenced HIV viral load, as well as HIV and CD4 specific immunity.

DETAILED DESCRIPTION:
The study will be based on forty HIV infected patients, receiving anti retroviral treatment (HAART), with CD4 levels between 150-350 and HIV plasma viral load < 5000, for at least 12 months and despite continuous anti-retroviral treatment. The patients will be randomly divided into two groups, one that will get the T cell vaccination, and the other that will serve as controls. The T cell vaccine will be prepared from autologous T cells that responded by specific proliferation to recombinant CD4, further expanded in vitro by IL-2, and then fixed by glutaraldehyde. Each vaccine portion will consist of 10,000 such cells suspended in saline and given subcutaneously every three months during the first year of the trial. The outcome measures will be CD4 levels, specific immunity to HIV antigens, immune activation profile and HIV plasma viral loads, determined sequentially during the 24 months of the trial. These outcome measures will be compared between the experimental and the control groups, to determine if this mode of treatment is effective in influencing CD4 levels as an additional mode of treatment during HIV infection.

ELIGIBILITY:
Inclusion Criteria:

1. CD4 cell counts -from 150 to 450/mm3 and stable for at least 12 months, and treatment with HAART for at least 6 months.
2. Positive cell proliferation assay to CD4 molecule
3. Low HIV viral load (<400 - 5000 copies/ml) for at least 12 months
4. No change of antiretroviral treatment for at least 6 months
5. Signed informed consent

Exclusion Criteria:

1. Concomitant immunosuppressive or antineoplastic treatment as well as chronic systemic glucocorticoid therapy.
2. Pregnancy and women without any efficacious contraception.
3. Clinically relevant liver disease (AST and/or ALT >2,5x upper limit of normal range, or total bilirubin > 3,5 mg/dl).
4. Serum creatinine >1,8mg/dl or creatinine clearance <30ml/min.
5. Patients who cannot fully understand the treatment protocol or are unable to sign the informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
CD4 T cell levels | one year follow up
HIV plasma viral load | one year follow up
Clinical HIV infection | one year follow up

SECONDARY OUTCOMES:
HIV specific immune responses | One year follow up
CD4 specific responses | One year follow up
Immune profile | One year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Klaris Riesenberg, M.D., Study Director — Soroka U Medical Center
Locations (1):
- Soroka Medical Center, Beersheba, Israel

REFERENCES:
- [Result] Abulafia-Lapid R, Bentwich Z, Keren-Zur Y, Cohen IR, Atlan H. T-cell vaccination against anti-CD4 autoimmunity in HIV-1 infected patients. J Clin Virol. 2004 Dec;31 Suppl 1:S48-54. doi: 10.1016/j.jcv.2004.09.017. PMID 15567094
- [Result] Abulafia-Lapid R, Mayan S, Bentwich Z, Keren-Zur Y, Avbramovitz Y, Cohen IR, Atlan H. T-cell vaccination against anti-CD4 autoimmunity in HIV-1 subtypes B and C-infected patients--an extended open trial. Vaccine. 2005 Mar 18;23(17-18):2149-53. doi: 10.1016/j.vaccine.2005.01.054. PMID 15755585